CLINICAL TRIAL: NCT00629785
Title: The Analysis of BMI, Asthma Prevalence, and Lung Functions of Schoolchildren in Southern Taiwan
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Other Study IDs: KMUH-IRB-960129
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2007-03

CONDITIONS: Asthma; Obesity
Keywords: asthma; pulmonary function tests; obesity
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The prevalence of obesity and asthma has increased in recent decades. We investigated the relationship between body mass index (BMI) and lung function, and also tried to determine if asthma prevalence differs between obese and non-obese children. We propose this cross-sectional, retrospective analysis to figure out whether the BMI is associated with elevated prevalence of asthma, and how their lung function changes in different BMI groups.

ELIGIBILITY:
Inclusion Criteria:

* students representing all grades in a total of 123 junior high schools in southern Taiwan (Kaohsiung and Pintong) between 1995-1996

Exclusion Criteria:

* failure to obtain ISAAC questionnaire
* failure to preform lung functions study

Ages: 13 Years to 16 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Chin Ko, Study Chair — Faculty of Public Health, Institute of Medicine, Kaohsiung Medical University, Kaohsiung, Taiwan